CLINICAL TRIAL: NCT03297138
Title: Fistula Laser Closure
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: FILAC
Record Dates: First submitted 2017-09-25; First posted 2017-09-29 (Actual); Last update posted 2018-05-30 (Actual); Status verified 2018-05

CONDITIONS: Fistula;Rectal
MeSH Terms: conditions — Rectal Fistula

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: FiLAC laser — The technique consists in applying in a radial way to 360 ° an energy laser in the fistulous route. This energy allows a thermal destruction by coagulation of the wall of the fistula and the fabrics of granulations in a circular and regular way as well as a shrinkage of neighbouring fabrics. The repair is made by a call of macrophages and fibroblasts of neighbouring healthy fabrics so ending in a closure of the fistulous route

SUMMARY:
The anal complex fistula constitutes a challenge in proctologic surgery because of the of its therapeutic care complexity due to the frequency of recurrences and the necessity to protect the sphincter function.

For several years,differents techniques were developed "said sphincter sparing techniques" to handle fistulas at risk on the anal continence.

Recently there is one of them , named FiLAC using a clip system not yet evaluated.

The purpose is to assess the success rate of his new surgery technique.

ELIGIBILITY:
Inclusion Criteria:

* Patient with anal fistula drained at least 3 months before inclusion.

Exclusion Criteria:

* Fistula not well drained

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient having a surgical indication using FiLAC laser technique
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2016-09-16 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
surgery success rate | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: Undecided